CLINICAL TRIAL: NCT06207513
Title: Single-used Versus MultiPlE-used Endotracheal suCtIon cAtheters in Mechanically ventiLated ICU Patients: the SPECIAL-ICU Trial
Brief Title: Single-used Versus MultiPlE-used Endotracheal suCtIon cAtheters in Mechanically ventiLated ICU Patients
Acronym: SPECIAL-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4112023
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-06

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention I group (Experimental): Patient intubated with an endotracheal tube and on a mechanical ventilator will receive endotracheal suctioning procedure using a single-used open endotracheal suction catheter that is used only for one-time suctioning attempt and discarded after each endotracheal suction cycle. A new catheter will be used for each endotracheal suctioning procedure.
  Interventions: Procedure: Suction Circuit Flushing with Chlorhexidine
- Intervention II group (Experimental): Patient intubated with an endotracheal tube and on a mechanical ventilator will receive endotracheal suctioning procedure using an open endotracheal suction catheter that is used multiple times during a 12-hour nursing shift. Flushing of the suctioning circuit will be performed with 40 ml of chlorhexidine gluconate 0.2% after every endotracheal suction procedure
  Interventions: Procedure: Suction Circuit Flushing with Chlorhexidine
- Control group (Other): Patients intubated with an endotracheal tube and on a mechanical ventilator will receive standard care. This is the endotracheal suctioning procedure using an open endotracheal suction catheter that is used multiple times during a 12-hour nursing shift. Flushing of the suctioning circuit is standardised performed using normal saline after every endotracheal suction procedure.
  Interventions: Procedure: Suction Circuit Flushing with Chlorhexidine

INTERVENTIONS:
Procedure: Suction Circuit Flushing with Chlorhexidine — Patient intubated with an endotracheal tube and on a mechanical ventilator will receive endotracheal suctioning procedure using an open endotracheal suction catheter that is used multiple times during a 12-hour nursing shift. Flushing of the suctioning circuit will be performed with 40 ml of chlorhexidine gluconate 0.2% after every endotracheal suction procedure

SUMMARY:
In low and middle-income countries, open endotracheal suction catheters are used multiple times to perform suctioning due to limited resources [1,2]. Currently, there is limited evidence for using a new suction catheter for each suction pass, acknowledged in a review article of endotracheal suction procedures in paediatric populations [3]. Additionally, the latest artificial airway suctioning practice guidelines published by the American Association for Respiratory Care in 2022 did not mention any recommendations regarding suction catheter changing frequency [4]. The guidelines adopted a study conducted in 2001 which showed that reusing an open tracheal suctioning catheter is safe and cost effective [5]. Therefore, the current evidence of reusing suctioning catheters remains unclear, which rationalize the reason why some resource limited Intensive Care Units (ICUs) use the catheter multiple times during a 12-hour shift, and possibly explain the high ventilator associated pneumonia (VAP) incidence in these ICUs [1,2].

Therefore, this feasibility study will propose to explore whether single-used suction catheters or multiple used open endotracheal tracheal suctioning catheters flushed with chlorhexidine are associated with reduced VAP incidence and its impact on mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥ 18 years old) who are admitted to the ICU, intubated with an endotracheal tube and receiving mechanical ventilation support directly after intubation with an expected mechanical ventilation support of at least 48 hours.
* All adults' patients meeting the above criteria whose relatives agree for them to be part of the study via deferred consent process

Exclusion Criteria:

* Patients who have received already standard care at ICU admission (the use of an endotracheal suction catheter multiple times during endotracheal suction procedures)
* Patients with contraindications to endotracheal suctioning procedure such as increased intracranial pressure, severe haemoptysis, and cerebrospinal fluid leaks.
* Patients who are previously intubated during the current hospital admission.
* Patients expected to receive mechanical ventilation less than 72 hours.
* Patients diagnosed with pneumonia at ICU admission.
* Patients having a Modified Clinical Pulmonary Infection Score (MCPIS) of 5 or greater.
* Patients with atelectasis, ARDS, and pulmonary oedema.
* Patients known to be allergic to chlorhexidine.
* Patients whose family (next-of-kin) have not provided deferred consent within 48 hours after ICU admission will be excluded and standard care will be provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | through study completion, an average of 1 year
  The feasibility and acceptability of the proposed intervention among healthcare professionals in study settings and determine methods for the design of a conclusive randomized controlled trial.

SECONDARY OUTCOMES:
Patients outcome | through study completion, an average of 1 year
  Will measure the impact of the proposed intervention on mechanically patients outcomes including Ventilator associated pneumonia incidence (using the modified clinical pulmonary infection score) and length of ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dkahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eid MH, Hambridge K, Schofield P, Latour JM. Single-Use Versus Multiple-Use Endotracheal Suction Catheters in Mechanically Ventilated Patients: A Feasibility Randomised Controlled Trial. Nurs Crit Care. 2026 Jan;31(1):e70237. doi: 10.1111/nicc.70237. PMID 41501433

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT06207513/SAP_000.pdf
  • Informed Consent Form (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT06207513/ICF_001.pdf